CLINICAL TRIAL: NCT06788678
Title: A Randomized Controlled Trial of a Web-Based Moral Elevation Intervention for Veterans With PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D5081-R
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Web-Based Intervention; Veterans; Randomized Controlled Trial; Moral Elevation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either the MOVED condition (target intervention) or a Supportive Care Control (SCC) condition. Both conditions are accessed through an online portal. The MOVED condition includes the moral elevation treatment with intervention content and goal setting activities. The SCC condition is a present-centered, nondirective interaction that aims to control for the nonspecific therapeutic effects of engaging in regular web-based session. Specifically, it includes psychoeducation materials about PTSD symptoms, functioning, and resources for related stressors. Key intervention components of MOVED (e.g., moral elevation exercises and goal-setting) will be excluded from SCC.
Who Masked: Outcomes Assessor
Masking Description: All staff conducting baseline and follow-up assessments (i.e., posttreatment, 3-months, 6-months) will be blinded to the assigned condition for all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MOVED (Experimental): Moral Elevation Online Intervention for Veterans Experiencing Distress.
  Interventions: Behavioral: MOVED
- Supportive Care Control (Active Comparator): Present-centered, nondirective intervention
  Interventions: Other: Supportive Care Control

INTERVENTIONS:
Behavioral: MOVED — MOVED includes 8 self-guided, web-based sessions administered over 4 weeks. Web-based sessions include 3 core components: (1) elicit moral elevation, (2) engage in reflection about moral elevation response, and (3) set a behavioral goal that is inspired by the moral elevation exercise.
  Other Names: Moral Elevation Online Intervention for Veterans Experiencing Distress
  Arms: MOVED
Other: Supportive Care Control — A present-centered, nondirective intervention that aims to control for the nonspecific therapeutic effects of supportive care. In this case, the effects of engaging in regular web-based sessions that convey information about PTSD symptoms. Sessions will include psychoeducation materials about PTSD symptoms, functioning, and resources for dealing with related stressors. Key components of MOVED will be strictly excluded.
  Arms: Supportive Care Control

SUMMARY:
Despite the availability of evidence-based treatments for PTSD, there are many challenges to successful trauma recovery for Veterans including difficulties starting and completing these treatments and gaps in fully addressing additional important treatment targets including lower social functioning and quality of life. Alternative, stand-alone treatment options that address a range of outcomes and can be easily accessed are needed to expand the reach of PTSD treatment to Veterans. One way to address this need is with a positive psychology intervention called MOVED, which has shown promise in a prior pilot study. MOVED is a web-based, self-guided intervention (8 sessions, 4 weeks) that uses moral elevation-feeling inspired by others' virtuous actions. This clinical trial will test if MOVED leads to decreased PTSD symptoms and increased social functioning and quality of life compared to a generic supportive treatment that does not focus on moral elevation. Results will help determine if MOVED is a useful alternative approach to target trauma recovery among Veterans with PTSD.

DETAILED DESCRIPTION:
Poor treatment engagement and retention with evidence-based practices (EBPs) are significant problems for Veterans with posttraumatic stress disorder (PTSD). Additionally, Veterans with PTSD also face significant issues with impaired social functioning and diminished quality of life; however, research suggests EBPs may not full address these other important treatment targets despite their ability to reduce PTSD symptoms. These limitations showcase how difficult it is to successfully treat PTSD and highlight the need for novel, stand-alone approaches as alternatives to current treatments that can further facilitate trauma recovery. Accessible and easily disseminated treatments are needed to target ongoing concerns for Veterans including PTSD symptoms, lower QOL, and poor social functioning. One approach that is well-suited to target these issues is a positive psychology-based intervention that focuses on eliciting moral elevation and its benefits. Moral elevation is a positive, emotional state of feeling inspired or moved by witnessing others' virtuous actions, which leads to greater social engagement and self-improvement motives. Moral Elevation Online Intervention for Veterans Experiencing Distress (MOVED) was previously developed as a web-based, self-guided intervention (8 sessions; 4 weeks) and piloted with a sample of Veterans experiencing significant PTSD symptoms and moral injury-related distress. Results from the VA funded pilot trial suggested MOVED was highly feasible and acceptable by Veterans, it demonstrated high levels of treatment engagement, and Veterans reported positive treatment outcomes including large decreases in PTSD symptoms and medium increases in quality of life. Given the promising findings from the MOVED pilot trial, the goal of this proposed study is to proceed with the next phase of treatment development for MOVED by conducting a powered efficacy trial with a sample of Veterans diagnosed with PTSD for at least one year. Following recent adaptations to MOVED that were informed by Veteran feedback from the pilot trial and with input from key stakeholders (researchers, clinicians, and Veterans with PTSD), a refined version of MOVED will be examined with a randomized controlled trial (RCT). This RCT will test the efficacy of MOVED compared to a supportive care control treatment in decreasing PTSD symptom severity, increasing social functioning, and increasing quality of life. The targeted sample will include 250 Veterans who have a PTSD diagnosis for at least one year. Eligible participants will be randomized to the MOVED condition or a supportive care control condition. Both interventions will be self-guided, web-based, and will include 8 sessions lasting 4 weeks. The supportive care control treatment will be a present-centered, nondirective intervention that aims to control for the nonspecific therapeutic effects of supportive care, whereas MOVED will focus on eliciting experiences of moral elevation, guided reflection of those experiences, and facilitating the pursuit of weekly behavioral goals related to experiences of elevation. All participants in both conditions will complete clinician-administered interviews and self-report measures to assess outcomes at baseline, posttreatment, 3-month, and 6-month follow-up. Additionally, potential mechanisms of action on treatment outcomes will be assessed at each session including experiences of moral elevation and treatment adherence. Results from this study will indicate whether MOVED is a viable treatment that can reduce PTSD symptoms, boost quality of life, and enhance social functioning; thus, expanding the number of treatment options available for PTSD care.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a VISN 17 health care system
* English-speaking and able to provide written informed consent
* Willingness to complete study procedures and be randomized
* Internet access and an electronic device to complete the web-based sessions
* Current diagnosis of PTSD based on the CAPS-5
* History of PTSD diagnosis for at least 1 year

Exclusion Criteria:

* History of severe traumatic brain injury indicated by medical record review and the Ohio State Traumatic Brain Injury Identification Method (OSU TBI-ID)
* Current psychosis or mania as indicated by medical record review and the Mini International Neuropsychiatric Interview (MINI)
* Current suicide risk based on the Beck Depression Inventory-II (BDI-II)
* Currently enrolled and actively participating in a trauma-focused treatment including:

  * Cognitive Processing Therapy
  * Prolonged Exposure
  * Eye Movement Desensitization Reprocessing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | Follow-up assessments at posttreatment, 3-months, and 6-months.
  The CAPS-5 is a 30-item structured interview that will be used to assess clinician-rated PTSD symptom severity (range = 0-80).
World Health Organization Quality of Life - Brief Version (WHOQOL-BREF) | Follow-up assessments at posttreatment, 3-months, and 6-months.
  The WHOQOL-BREF is a 26-item self-report measure that will be used to assess overall quality of life with 4 domains (physical health, psychological health, social relationships, and environment). Subscales scores are computed by summing all items for each subscale, then all scores are transformed to a range of 0-100. A higher score signifies higher or better quality of life.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Follow-up assessments at posttreatment, 3-months, and 6-months.
  The WHODAS 2.0 is a self-report measures of functioning. Two socially-oriented subscales comprised of 13 items total will be used to assess social functioning across the Getting Along and Participation domains. Higher scores indicate greater functioning.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Follow-up assessments at posttreatment, 3-months, and 6-months.
  The PCL-5 is a 20-item self-report measure that will be used to assess PTSD symptom severity (range 0 = 80). Higher scores indicate greater symptom severity.
Moral Injury and Distress Scale (MIDS) | Follow-up assessments at posttreatment, 3-months, and 6-months.
  The MIDS is a 24-item self report measure that will be used to assess moral injury distress (range = 0-72). Higher scores indicate greater distress.
Engagement with Beauty Scale (EBS) - Moral Beauty Subscale | Follow-up assessments at posttreatment, 3-months, and 6-months.
  The EBS is a self-report measure that will be used to assess engagement with moral beauty or trait-level moral elevation. The moral beauty subscale includes 7 items (range = 6-42). Higher scores indicate greater engagement with moral beauty.
Purpose in Life - Short Form (PIL-SF) | Follow-up assessments at posttreatment, 3-months, and 6-months.
  The PIL-SF is a 4-item self-report measure that will be used to assess perceived meaning and purpose in life (range = 4-28). Higher scores indicate greater purpose in life.
Posttraumatic Growth Inventory (PTGI) | Follow-up assessments at posttreatment, 3-months, and 6-months.
  The PTGI is a 21-item self-report measure that will be used to assess posttraumatic growth (range = 0-105). Higher scores indicate greater posttraumatic growth.

OTHER OUTCOMES:
State Moral Elevation Scale (SMES) | Administered during 8 sessions across 4 weeks
  The SMES is a 9-item self-report measure that will be used to assess state-level moral elevation experienced during each session for both conditions (range = 0-36). Higher scores indicate greater moral elevation.

CONTACTS AND LOCATIONS:
Overall Officials: Adam P. McGuire, PhD, Principal Investigator — Central Texas Veterans Health Care System, Temple, TX
Locations (1):
- Central Texas Veterans Health Care System, Temple, TX, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared pursuant to a Data Use Agreement (DUA).
Time Frame: 1 year after publication